CLINICAL TRIAL: NCT04840472
Title: Pilot Evaluating 111In-Panitumumab for Nodal Staging in Head and Neck Cancer
Brief Title: Study Evaluating 111In-Panitumumab for Nodal Staging in Head and Neck Cancer
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: tentatively suspended until drug manufacturing is available
Sponsor: Stanford University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-58398; ENT0083 (Other: OnCore); NCI-2021-05694 (Registry Identifier: National Cancer Institute: Clinical Trials Reporting Program)
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 111-In panitumumab (Experimental): The study drug (111In panitumumab) 5 mCi, allowable range 4.5 to 5.5 will be administered on Day 0, and subjects will undergo one 111In panitumumab SPECT/CT imaging anytime between Day 1 and Day of Surgery. Subjects will undergo surgical resection after infusion of 111In panitumumab.
  Interventions: Drug: 111I-n panitumumab; Procedure: Single photon emission computed tomography/computed tomography (SPECT/CT) scans

INTERVENTIONS:
Drug: 111I-n panitumumab — Imaging Agent
Procedure: Single photon emission computed tomography/computed tomography (SPECT/CT) scans — Day 1 to 5 (Day of Surgery inclusive)

SUMMARY:
The primary purpose of the study is to assess the safety of 111In-panitumumab as a molecular imaging agent in patients with Head and Neck Squamous Cell Carcinoma.

The secondary objective is to compare sensitivity and specificity of identifying sentinel lymph nodes by systemic injection of 111In-panitumumab prior to Day of Surgery versus conventional local injection with an optical dye at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed diagnosis of squamous cell carcinoma of the head and neck.
* Subjects diagnosed with any T stage, any subsite within the head and neck that are scheduled to undergo surgical resection. Subjects with recurrent disease or a new primary will be allowed.
* Planned standard of care elective neck dissection for a cN0 or cN1 disease. Clinical N1 disease will be defined as metastasis in a single, ipsilateral lymph node, 3 cm or less in greatest dimension by clinical exam, cross sectional imaging or metabolic imaging.
* Have acceptable hematologic status, coagulation status, kidney function, and liver function including the following clinical results:
* Hemoglobin ≥ 9 gm/dL
* White blood cell count > 3000/mm3
* Platelet count ≥ 100,000/mm3
* Serum creatinine ≤ 1.5 times upper reference range

Exclusion Criteria:

* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment.
* History of infusion reactions to monoclonal antibody therapies.
* Pregnant or breastfeeding.
* Magnesium or potassium lower than the normal institutional values.
* Subjects receiving Class IA (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents.
* Subjects with a history or evidence of interstitial pneumonitis or pulmonary fibrosis.
* Severe renal disease or anuria.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Assess the safety of 111In panitumumab as a molecular imaging agent in patients with HNSCC. | 15 days
  Number of CTCAE v5.0 Grade 2 or higher adverse events by Day 15 determined that are significant, definitely or probably related to 111In panitumumab. Safety data will be summarized by grade, severity, and type.

SECONDARY OUTCOMES:
Compare sensitivity of systemic 111In panitumumab versus conventional local optical dye | 10 days after surgery
  Sensitivity of systemic 111In panitumumab of identifying sentinel lymph nodes versus sensitivity of conventional local optical dye in identifying sentinel lymph nodes using histopathology will be compared
Compare specificity of systemic 111In panitumumab versus conventional local optical dye | 10 days after surgery
  Specificity of systemic 111In panitumumab of identifying sentinel lymph nodes versus specificity of conventional local optical dye in identifying sentinel lymph nodes using histopathology will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Fred Baik, MD, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No